CLINICAL TRIAL: NCT01910688
Title: Use of Endoscopically Delivered Radiofrequency Ablation for the Treatment of Ptients Who Have Undergone Roux-en-Y Gastric Bypass and Have Failed to Achieve/ Maintain Satisfactory Excess Body Weight Loss
Brief Title: Use of Radiofrequency Ablation for RGB Salvage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-600
Record Dates: First submitted 2013-07-24; First posted 2013-07-30 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Obesity
Keywords: RGB Salvage, RFA
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RFA treatment (Radiofrequency ablation) (Experimental): If eligible for enrollment, patients receive initial RFA treatment at 0 month. Patients return to the study site at 3.5 months to review weight data since initial RFA. If the patient has not reached ideal body weight, the patient is scheduled for endoscopy with RFA at 4 months. All patients are seen at 7.5months and if the patient has not reached ideal body weight, the patient is scheduled for endoscopy with RFA at 8 months. All patients are seen at the study site at 12 months for final clinic weight.
  Interventions: Device: RFA treatment

INTERVENTIONS:
Device: RFA treatment — If eligible for enrollment, a focal ablation device is selected as an intervention(size according to physician preference) and mounted on the end of the endoscope and introduced via the mouth into the esophagus and gastric pouch. The gastric pouch is treated from the top of the gastric folds to and just through the stomal anastomosis.
  Other Names: HALO60, HALO90, HALO90 Ultra

SUMMARY:
The present study will assess the feasibility of using endoscopic radiofrequency ablation (RFA) to treat the gastric pouch and stoma with the intent to cause tissue contraction and decreased compliance after a failed Roux-en-Y gastric bypass.

DETAILED DESCRIPTION:
Obesity is a leading cause of preventable death in the United States, with approximately 300,000 related deaths per year. The most commonly performed bariatric surgical interventions are Roux-en Y gastric bypass (RGB) and laparoscopic adjustable gastric band placement. Despite the overall initial success of RGB to induce significant EBWL in the majority of patients, significant weight regain occurs in about 25% of patients at 2+ years following surgery. Given the preliminary success of endoscopic, non-surgical salvage interventions for the failed (uncomplicated) RGB patient, the present study will assess the feasibility of using endoscopic radiofrequency ablation (RFA) to treat the gastric pouch and stoma with the intent to cause tissue contraction and decreased compliance. A reduction of size and compliance may, as others have reported, result in re-establish weight loss and achieve an acceptable EBWL with minimal patient morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. History of RGB surgery at least 1 year prior to enrollment
2. Achievement of > 40% EBWL after RGB
3. Weight regain of > 25% of the lost weight at the time of enrollment. For example, if excess body weight was 50 kg prior to RGB, patient must have lost at least 20 kg after RGB, then regained at least 5 kg to be eligible for the present study
4. Age 18-70 inclusive
5. Subject is able to tolerate endoscopy and sedation
6. Subject agrees to participate, fully understands content of the informed consent, and signs the informed consent form (ICF)

Exclusion Criteria:

1. History of any bariatric surgery other than RGB, including lap band
2. History or presence of a gastrogastric fistula or gastric pouch / jejunal ulceration
3. Gastrojejunostomy > 4 cm in diameter (size estimated at time of endoscopy)
4. Perceived inability of the patient by the Investigator to comply with a post-treatment diet or medication regimen
5. History of alcohol, tobacco and/or controlled substance dependency that would impair the patient from complying with protocol requirements
6. Pregnancy
7. Subject is unable to provide informed consent for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Abrams, MD, Principal Investigator — Columbia University; Richard Rothstein, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia Univeristy, New York, New York

REFERENCES:
- [Derived] Abrams JA, Komanduri S, Shaheen NJ, Wang Z, Rothstein RI. Radiofrequency ablation for the treatment of weight regain after Roux-en-Y gastric bypass surgery. Gastrointest Endosc. 2018 Jan;87(1):275-279.e2. doi: 10.1016/j.gie.2017.06.030. Epub 2017 Jul 13. PMID 28713063

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RFA Treatment (Radiofrequency Ablation)
Started | 25
3.5month | 25
2nd RFA Treatment | 22
7.5months | 24
3rd RFA Treatment | 18
12months | 22
Completed | 20
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Patient who had undergone RGB at least 1 year prior to enrollment, achieved > 40% EBWL after surgery, and then regained > 25% of the lost weight.
Arm/Group | RFA Treatment (Radiofrequency Ablation)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Excess Body Weight Loss After RFA Treatment
Description: EBWL 12 months after enrollment
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of EBWL
Arm/Group | RFA Treatment (Radiofrequency Ablation)
Number analyzed (Participants) | 22
percentage of EBWL | 28.36 (28.830)

2. Secondary Outcome: Technical Feasibility: Percentage of Participants Who Completed RFA Treatment
Description: Technical feasibility of applying RFA to gastric pouch and gastrojejunostomy. This will be assessed by asking the physician for feedback on ease of use, ease of intubation and extubation,did the physician achieve tissue contact in targeted areas, was targeted area successfully ablated.
Time Frame: Day 0, month 4, month 8
Population: At 0 month, 25 received 1st RFA treatment; at 4 month, 22 received 2nd RFA treatment; at 8 month, 18 received RFA Treatment
Measure: Number; unit: percentage of participants
Arm/Group | RFA Treatment (Radiofrequency Ablation)
Number analyzed (Participants) | 25
percentage of participants
  Day 0 | 84
  Month 4 | 95.45
  Month 8 | 94.44

3. Secondary Outcome: Patient Tolerability
Description: Patient tolerability of the procedure. Patient tolerability will be measured by assessing adverse events related to the device or procedure. The Investigator will assess each adverse event with respect to severity and relationship to the study device.
Time Frame: 12 months
Measure: Number; unit: number of events
Arm/Group | RFA Treatment (Radiofrequency Ablation)
Number analyzed (Participants) | 25
number of events | 12

4. Secondary Outcome: Adverse Events
Description: Adverse event profile: Relationship to study device : Definite, Probable, Possible
Time Frame: 12 months
Measure: Number; unit: number of events
Arm/Group | RFA Treatment (Radiofrequency Ablation)
Number analyzed (Participants) | 25
number of events
  Definite | 6
  Possible | 2
  Probable | 3

ADVERSE EVENTS:
Arm/Group | RFA Treatment (Radiofrequency Ablation)
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RFA Treatment (Radiofrequency Ablation) (N=25)
GI bleed (Injury, poisoning and procedural complications) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RFA Treatment (Radiofrequency Ablation) (N=25)
Dysphagia (Injury, poisoning and procedural complications) | 2 (2)
Mucosal Bleeding (Injury, poisoning and procedural complications) | 2 (2)
Fever (Injury, poisoning and procedural complications) | 1 (1)
Vomiting, Nausea (Injury, poisoning and procedural complications) | 4 (5)
Abdominal tenderness. Oesophageal pain (Injury, poisoning and procedural complications) | 2 (3)
Fatigue (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less